CLINICAL TRIAL: NCT00491049
Title: Phase 4 Study on Effectiveness of Topical 0.5% Levofloxacin on Reduction of Preoperative Conjunctival Flora in Patients Scheduled for Intraocular Surgery
Brief Title: Effectiveness of Topical 0.5% Levofloxacin to Reduce the Conjunctival Bacterial Flora Before Intraocular Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Santen Gmbh (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LevoProMUC03
Record Dates: First submitted 2007-06-21; First posted 2007-06-25 (Estimated); Last update posted 2007-06-25 (Estimated); Status verified 2007-06

CONDITIONS: Conjunctival Bacterial Flora
Keywords: prophylaxis; intraocular surgery; endophthalmitis; antibiotic
MeSH Terms: conditions — Endophthalmitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 0.5% levofloxacin eye drops

SUMMARY:
The purpose of this study is to determine whether additional topical application of 0.5% levofloxacin is more effective in reducing the load of the conjunctival bacterial flora in patients scheduled for intraocular surgery than preoperative irrigation of the conjunctiva with povidone iodine alone.

DETAILED DESCRIPTION:
Endophthalmitis is serious complication of intraocular surgery. Previous studies have shown that the most common sources of bacteria causing endophthalmitis are the patients eyelid and conjunctival bacteria. [1, 2] The risk of postoperative endophthalmitis may be reduced by eliminating bacteria from the ocular surface at the time of the surgery.

The current standard for endophthalmitis prophylaxis at Ludwig-Maximilians-University in Munich, Germany is the irrigation of the conjunctival fornices with 1% povidone-iodine (PVI) prior to surgery. In general, patients do not receive topical antibiotic prior to surgery.

Ta and co-workers have demonstrated that a three-day application of topical ofloxacin resulted in less conjunctival cultures obtained before and after surgery compared to an application of antibiotic given one hour prior to surgery.[3] Furthermore, the same research group showed that the contamination rate of the microsurgical knives used during surgery decreased from 26% to 5% (P = 0.028) with a three day application of ofloxacin compared to a one-hour application.[4] The goal of the current proposal is to determine if we can improve on the current standard of endophthalmitis prophylaxis at Ludwig-Maximilians-University by using topical 5% levofloxacin prior to surgery. Given that the rate of endophthalmitis is quite low, we will use conjunctival bacterial flora and anterior chamber aqueous contamination rate as surrogate markers to determine the effectiveness of topical levofloxacin in reducing or eliminating bacteria from the ocular surface at the time of the surgery. The results of this prospective-randomized control trial may radically change the current practice of endophthalmitis prophylaxis, and levofloxacin may play a critical role in preventing postoperative endophthalmitis.

Study Protocol:

One hundred and forty patients will be randomized to control group and a study group:

* Control group: no antibiotic (70 patients). Standard protocol at the Department of Ophthalmology, Munich.
* Study group I: topical 0.5% levofloxacin four times per day for one day prior to surgery. In addition, one drop of topical levofloxacin is given three times with five minutes intervals, one hour prior to surgery (70 patients).

Five minutes prior to surgery both groups will receive topical povidone-iodine (10%) to scrub the periorbital area and 1% PVI to irrigate the conjunctiva (standard protocol). Patients will be draped in a sterile fashion and surgery will be initiated.

Conjunctival cultures for aerobic and anaerobic bacteria will be obtained at the following time-points:

• T0: (Baseline) at the day of the first interview (one week before surgery), prior to any application of antibiotic or povidone-iodine. Samples will be taken from both conjunctivas.

* T1: On the morning of the surgery, but prior to final treatment during the last hour before surgery. At this time, patients in both study groups will have received topical levofloxacin (one day and three days before surgery) treatment; patients in the control group will not have received any treatment with antibiotic. Samples will be taken also from both conjunctiva.
* T2: Immediately before surgery, 5-10 min after PVI scrub and PVI irrigation for both the control and study group, but only on the conjunctiva of surgery eye. In addition of sample of anterior chamber aqueous fluid is taken from the surgery eye by the responsible surgeon.
* T3: At the conclusion of surgery, again from the conjunctiva and the anterior chamber fluid of the surgery eye.

At every step, samples are taken from the conjunctiva with a standard dissolving Ca-alginate swab (Sanofi-Pasteur, Germany). The moistened swab should be taken via one rotational swipe over the lower conjunctiva without touching the lid or eyelashes. Additionally anterior chamber aqueous fluid will be obtained immediately before and after surgery. The cannulas (2x) used for the aspiration will be cultured in a separate broth culture, too.

Inclusion criteria:

- Patients undergoing surgery for cataract, glaucoma or vitrectomy.

Exclusion criteria:

* Patients who report to be allergic to levofloxacin or iodine
* Patients on topical antibiotic within the last 30 days
* Patients with acute conjunctivitis, blepharitis or dacryocystitis
* Patients under age of 18 years

Summary:

The results of this study may revolutionize the standard of endophthalmitis prophylaxis. It could be that the application of topical levofloxacin 5%, four times a day for one or three days prior to surgery, significantly reduce or eliminate bacteria from the ocular surface. Hence, topical levofloxacin may have a critical role in preventing postoperative endophthalmitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery for cataract, glaucoma or vitrectomy

Exclusion Criteria:

* Patients who report to be allergic to levofloxacin or iodine
* Patients on topical antibiotic within the last 30 days
* Patients with acute conjunctivitis, blepharitis or dacryocystitis
* Patients under age of 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2004-09; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Rate of culture positive results in thioglycolate broth from conjunctival swabs at defined time points | maximum 7 days before surgery until conclusion of surgery

SECONDARY OUTCOMES:
Numbers of colony forming units (CFUs) found on solid media. Specimens were cultured aerobically and micro-aerobically on blood agar plates and anaerobically on chocolate agar plates and CFUs were determined on each plate using a magnifying glass. | maximum 7 days before surgery until concluison of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Herminia Mino de Kapsar, PhD, Principal Investigator — Augenklinik der LMU
Locations (1):
- Augenklinik der LMU, Munich, Bavaria, Germany

REFERENCES:
- [Background] Speaker MG, Milch FA, Shah MK, Eisner W, Kreiswirth BN. Role of external bacterial flora in the pathogenesis of acute postoperative endophthalmitis. Ophthalmology. 1991 May;98(5):639-49; discussion 650. doi: 10.1016/s0161-6420(91)32239-5. PMID 2062496
- [Background] Bannerman TL, Rhoden DL, McAllister SK, Miller JM, Wilson LA. The source of coagulase-negative staphylococci in the Endophthalmitis Vitrectomy Study. A comparison of eyelid and intraocular isolates using pulsed-field gel electrophoresis. Arch Ophthalmol. 1997 Mar;115(3):357-61. doi: 10.1001/archopht.1997.01100150359008. PMID 9076208
- [Background] Ta CN, Egbert PR, Singh K, Shriver EM, Blumenkranz MS, Mino De Kaspar H. Prospective randomized comparison of 3-day versus 1-hour preoperative ofloxacin prophylaxis for cataract surgery. Ophthalmology. 2002 Nov;109(11):2036-40; discussion 2040-1. doi: 10.1016/s0161-6420(02)01236-8. PMID 12414411
- [Background] De Kaspar HM, Chang RT, Shriver EM, Singh K, Egbert PR, Blumenkranz MS, Ta CN. Three-day application of topical ofloxacin reduces the contamination rate of microsurgical knives in cataract surgery: a prospective randomized study. Ophthalmology. 2004 Jul;111(7):1352-5. doi: 10.1016/j.ophtha.2003.10.032. PMID 15234136
- [Background] Mino de Kaspar H, Chang RT, Singh K, Egbert PR, Blumenkranz MS, Ta CN. Prospective randomized comparison of 2 different methods of 5% povidone-iodine applications for anterior segment intraocular surgery. Arch Ophthalmol. 2005 Feb;123(2):161-5. doi: 10.1001/archopht.123.2.161. PMID 15710810
- [Derived] Mino de Kaspar H, Kreutzer TC, Aguirre-Romo I, Ta CN, Dudichum J, Bayrhof M, Klauss V, Kampik A. A prospective randomized study to determine the efficacy of preoperative topical levofloxacin in reducing conjunctival bacterial flora. Am J Ophthalmol. 2008 Jan;145(1):136-142. doi: 10.1016/j.ajo.2007.08.031. Epub 2007 Nov 8. PMID 17996212
- See also: Website of the university eye hospital at the Ludwig-Maximilians University in Munich — http://augenklinikmuenchen.de